CLINICAL TRIAL: NCT02667015
Title: Development of an Anxiety Sensitivity-Based Intervention for Substance Use and Anxiety Comorbidity
Acronym: SUD/Anx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 126253
Record Dates: First submitted 2014-09-05; First posted 2016-01-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-01

CONDITIONS: Other (or Unknown) Substance Use Disorders
Keywords: Substance Use Disorders; Anxiety; Anxiety Sensitivity; Brief Intervention; Treatment
MeSH Terms: conditions — Substance-Related Disorders; Anxiety Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anxiety Sensitivity Intervention (Experimental): Group receives the 3-week, 6-session Anxiety Sensitivity Intervention. This is a 6-session psychotherapy occurring twice weekly (60-90 minutes) for three weeks. This psychotherapeutic treatment is focused on reducing anxiety sensitivity and includes many components, but primarily consists of psychoeducation about the relationship between anxiety and substance use disorders, interoceptive exposures, in vivo exposures, and cognitive challenging.
  Interventions: Behavioral: Psychotherapy (Anxiety Sensitivity Intervention)
- Control Group (No Intervention): Receives only treatment as usual

INTERVENTIONS:
Behavioral: Psychotherapy (Anxiety Sensitivity Intervention) — 3 week, 6-session psychotherapy targeting anxiety sensitivity
  Arms: Anxiety Sensitivity Intervention

SUMMARY:
The aim of the current study is to develop and pilot test an anxiety sensitivity-based intervention for co-occurring substance use disorders (SUDs) and anxiety. Research questions include determining whether a broadly-applicable AS-based intervention can significantly decrease both substance misuse and anxiety. Secondary aims include examining the impact of this intervention on general functioning and depressive/anxious symptoms. In phase I, an initial pilot was conducted to examine the feasibility, safety, and patient satisfaction with the protocol, and to estimate potential efficacy of the protocol. In phase II, participants will be randomized to the intervention or a control condition.

DETAILED DESCRIPTION:
The aim of the current study is to develop and pilot test an anxiety-sensitivity based intervention for co-occurring SUDs and anxiety. In the proposed study, the investigators will develop, refine, and pilot-test an innovative cognitive-behavioral therapy (CBT) for patients who suffer from substance use disorders as well as anxiety. The goal of the research group in the proposed study is to design a protocol that can be testable on a larger sample within an externally-funded, randomized controlled trial. The investigators plan to submit a proposal for this larger grant to the National Institute on Drug Abuse, as outlined in our external funding statement.

Research questions include determining whether a broadly-applicable anxiety sensitivity based intervention can significantly decrease both substance misuse and anxiety. Secondary aims include examining the impact of this intervention on general functioning and depressive/anxious symptoms. In this translational research project, strategies that have been demonstrated to impact the psychological mechanisms thought to underlie both illnesses will be tested in a "real world" clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* score higher than 25 (established clinical cutoff) on the Anxiety Sensitivity Index (ASI; Peterson & Plehn, 1999)
* meet the DSM diagnostic criteria for current substance abuse or psychological dependence

Exclusion Criteria:

* active psychosis, suicidality, mania, or current physiological withdrawal symptoms that necessitate medical detoxification; no substance use in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in total score on Anxiety Sensitivity Index (ASI; Peterson & Plehn, 1999), from baseline (pre-treatment) to ASI score at 3-months post-treatment. | Pre, Post, 3-month follow-up
  The ASI is a self-report measure consisting of 16 questions which ask about past-week fear of physical and psychological symptoms of anxiety and fear of potential sequelae of anxiety (e.g., "When I notice my heart is beating rapidly, I worry that might have a heart attack"; or "When my stomach is upset, I worry I might be seriously ill"). Scores over 25 are suggestive of clinically significant anxiety sensitivity (Peterson & Plehn, 1999).
Change in Percent Days Abstinent over the past 30 days on the Timeline Follow-Back (TLFB; Sobell & Sobell, 1996), from Pre-treatment to 3-months post-treatment. | Pre, Post, 3-Month Follow-Up (measure queries past 30 days only at these time points)
  The TLFB is an interview which asks patients to retrospectively report on daily drinking quantity and frequency for the past 30 days. Using a calendar, the interviewer asks the respondent to identify important holidays and other memorable events over the retrospective time window, and then uses these events to help cue the respondent's memory of alcohol /drug use quantity and frequency over this period. Using these prompts and the respondent's knowledge of his/her own drinking/drug use patterns, an report of types of drug used and estimates of quantity of use is obtained for each day in the window. In the current study, the baseline and follow-up TLFBs covered the past 90 days; the post-treatment TLFB covered the past 30 days.

SECONDARY OUTCOMES:
Change in total score on Depression, Anxiety, and Stress Scales (DASS; Brown, Chorpita, Korotitsch, & Barlow, 1997). | Pre, Post, 3-month Follow-up
  The DASS is a 21-item self-report questionnaire which provides total scores for anxiety, depression, and stress subscales. The Depression scale assesses symptoms of dysphoria, hopelessness, devaluation of life, self-deprecation, anhedonia, lack of interest/involvement, and inertia. The Anxiety scale assesses symptoms of autonomic arousal, skeletal musculature effects, situational anxiety, and subjective experience of anxious affect. The Stress scale assesses symptoms of difficulty relaxing, nervous arousal, agitation, irritability/over-reactivity, and impatience. The DASS queries about symptoms in the past week and therefore outcome will be change in total score from pre-treatment to 3 months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Blaise l Worden, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States